CLINICAL TRIAL: NCT02021877
Title: Evidence Based Diagnostics and Treatment Planning Solution for Traumatic Brain Injuries - the TBIcare Project
Brief Title: Evidence Based Diagnostics and Treatment Planning Solution for Traumatic Brain Injuries
Status: Completed | Type: Observational
Sponsor: Turku University Hospital (Other Government)
Collaborators: Cambridge University Hospitals NHS Foundation Trust (Other); Imperial College London (Other); VTT Technical Research Centre of Finland (Other); GE Healthcare (Industry); Kaunas University of Technology (Other)
Responsible Party: Sponsor
Other Study IDs: EU funded project nr 270259
Record Dates: First submitted 2013-12-20; First posted 2013-12-27 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Traumatic Brain Injury
Keywords: Brain trauma; ICP measurement; cranial CT / MRI; Glasgow Coma Score; acute TBI; EEG; metabolic, proteomic, and genetic biomarkers of TBIs; injury mechanism
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum and plasma samples for proteomic, metabolomic and genetic analyses.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- TBI subjects: Unselected adult patients with acute TBI from the Emergency Departments of the recruiting hospitals
- Control subjects: Acute orthopaedic non-trivial trauma that needs either surgery or conservative measures and clinical follow-up (including mere superficial soft tissue injuries)

SUMMARY:
Adult patients, age ≥ 18 years, with clinically diagnosed mild, moderate or severe brain trauma will be asked to participate in the study. This prospective database will consist of 400 subjects with TBI, 200 from both TUCH and Cambridge Addenbrooke's Hospital. In addition, 100 controls will be recruited, with 50 from both centres.This study is a prospective clinical observational study with detailed data collecting. All patients will be treated according to the accepted, standardized, existing guidelines that are based on national and international recommendations. New treatment interventions will NOT be evaluated during the data acquisition for this study.

DETAILED DESCRIPTION:
Aim in this study is to collect large amounts of data in adult subject population, who have suffered mild, moderate or severe brain trauma. This data will be added up to the existing large TBI databases from IMPACT as well as to the retrospective brain trauma data sets collected at the Turku University Hospital after the year 1995 and to the prospectively collected existing data set from the University of Cambridge.

Data will contain patient characteristics, injury mechanisms, and patients' physiological status and findings immediately after the incident as well as through the processes of diagnostics, emergency treatment and in-hospital care. All data during these phases will follow the recommendations of Common Data Elements (advanced version) in TBI studies by the IMPACT investigators.

Immediate head CT will be performed according to the existing guidelines, and head MRI with modern techniques as soon as the patient's wellbeing will allow the imaging to be done.

During the intensive care unit (ICU) visit a database of EEG signals will be collected and the relevant information components will be extracted to provide inputs for the care decision algorithm. The aim is to investigate the feasibility of continuous EEG monitoring on the detection of epileptic seizures and other adverse events to enable rapid intervention during the patient's ICU stay and to improve outcome prediction.

The investigators will also search new metabolomic, lipidomic, and genetic biomarkers related to TBIs through analyzing blood samples drawn in different time points.

Based on all these factors, simulation models will be brought up as to help clinicians determine the earliest possible prognosis and to decide, whether patient would benefit from a particular care during the acute phase of a TBI.

ELIGIBILITY:
Inclusion Criteria:

* Severe or moderate brain trauma subjects with need of ICU care:
* Glasgow Coma Score (GCS) ≤ 8 after the primary stabilization has been performed in the field (= patient not hypoxic or hypotensive) and at least 30 min interval from the moment of injury.
* GCS 9 - 13 and the patient is deteriorating
* The patient has GCS ≤ 13 and has other injuries, which require interventions for hemodynamic or ventilatory incidents
* The patient is in urgent need of neurosurgery (craniotomy, impression skull fracture, severe haemorrhagic contusion, or ICP measurement)

Moderate or mild brain trauma not in need of ICU care:

- All other patients who fulfil the diagnostic criteria for an acute TBI but without any exclusion criteria defined below

Exclusion Criteria:

* Age < 18 years at study entry
* Blast-induced TBI
* Perforating or penetrating mechanism of TBI
* Unable to live independently because of a brain disease (= e.g. people with moderate dementia, Down's syndrome, cerebral palsy etc.) or other medical cause before the injury
* TBIs or suspected TBIs not needing cranial CT imaging (excludes the mildest TBIs with negligible risk for incomplete recovery)

Inclusion criteria for control subjects

* Age ≥ 18 years at study entry
* Acute orthopaedic non-trivial trauma that needs either surgery or conservative measures and clinical follow-up (including mere superficial soft tissue injuries)

Exclusion criteria for control subjects

* Age < 18 years at study entry
* Loss of consciousness or amnesia or neurological symptoms or signs in conjunction with the injury, or suspicion of such
* External injuries of the head caused by the acute injury
* Acute injury of the spinal column and/or cord (including whiplash-injuries of the neck) - superficial soft tissue injuries without neurological symptoms or signs are not an exclusion
* Any earlier TBI with loss of consciousness, amnesia or prolonged symptoms (days or more)
* Suspicion or signs of TBI (recent or remote) in brain MRI
* Trauma that needs care or observation at ICU, at any time point during the acute hospital period
* Previous neurological illnesses with obvious permanent alteration in CNS function (cerebral palsy, multiple sclerosis, stroke, encephalitis, degenerative CNS disorders, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients, age ≥ 18 years, with clinically diagnosed mild, moderate or severe brain trauma will be asked to participate in the study. If such possible subjects are either unconscious, sedated or confused to the extent, that no personal decisions can be drawn, her next of kin will be asked for the permission to include the subject in question to the study. Control group subjects will be patients with acute orthopaedic injuries without any signs of eventual concomitant brain trauma of any degree. The source populations will consist of citizens from the local catchment areas of the participating centres.
Sampling Method: Non-Probability Sample
Enrollment: 396 (Actual)
Dates: Start 2011-02; Primary Completion 2014-04 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Glasgow Outcome Scale -extended | Time for outcome assessment is nine months (range 3 to 12 months) from the injury.
  •General outcome is assessed using the Glasgow Outcome Scale, extended version (GOS-E)

SECONDARY OUTCOMES:
QOLIBRI | 3 - 12 months from injury
  •The quality of life is assessed using QOLIBRI
CANTAB | 3 - 12 months from injury
  •Cognitive outcome is assessed using CANTAB, an electronic test battery to evaluate neuropsychological function. The subtests used include tests of visual memory, executive function, working memory, planning, attention, semantic/verbal memory, decision-making, and response control
Rivermead Post Concussion Symptom Questionnaire | 3 - 12 months from injury
  •Subjective outcome is assessed using the Rivermead Post-Concussion Symptom Questionnaire (RPCSQ)
SF-36 | 3 - 12 months from injury
  •Subjective outcome is assessed using the SF-36 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Olli Tenovuo, MD, PhD,, Principal Investigator — Turku University Hospital
Locations (2):
- Turku University Hospital, Turku, Finland
- Cambridge Addenbrooke's Hospital, Cambridge, United Kingdom